CLINICAL TRIAL: NCT05608395
Title: 11C-methionine in Diagnostics and Management of Glioblastoma Multiforme With Rapid Early Progression Patients Prior to Adjuvant Oncological Therapy (GlioMET)
Brief Title: 11C-methionine in Diagnostics and Management of Glioblastoma Multiforme Patients (GlioMET)
Acronym: GlioMET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MOU-2020-01
Record Dates: First submitted 2021-02-25; First posted 2022-11-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma Multiforme
Keywords: rapid early progression; 11C-Methionine; MET-PET/CT
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: 11C-Methionine PET/CT Arm is to be compared to historical cohort A(hist.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 11C-Methionine PET/CT Arm (Experimental): The cohort consists of patients:
  * diagnosed with GB
  * with confirmed REP
  * indicated for adjuvant chemoradiotherapy
  * will undergo the 11C-MET PET/CT
  Interventions: Drug: 11C-Methionine PET/CT
- Arm A-historical (No Intervention): The cohort consists of a historical group of patients collected in the period 2014-2018:
  * with diagnosed GB
  * with confirmed REP
  * were indicated for adjuvant chemoradiotherapy

INTERVENTIONS:
Drug: 11C-Methionine PET/CT — 11C-Methionine PET/CT will be applied in patients in 11C-Methionine PET/CT Arm, based on planning MRI, prior chemo/radiotherapy (2 weeks prior C1D1)
  Other Names: Methionine application
  Arms: 11C-Methionine PET/CT Arm

SUMMARY:
Glioblastoma multiforme (GBM) is the most common primary brain cancer. The treatment of GBM consists of a combination of surgery and subsequent oncological therapy, i.e. radiotherapy, chemotherapy, or combination of both at te same time. If post-operative oncological therapy involves irradiation, magnetic resonance imaging (MRI) is planned. Unfortunately, in some cases, a very early worsening (progression) or return (recurrence) of the disease is observed several weeks after the surgery, i.e. rapid early progression (REP). Radiotherapy planning is based on this MRI in all patients. However, a subset of patients with REP have a less favorable prognosis with this treatment management. The investigators therefore assume that these patients need a more thorough examination to form a precise radiotherapy plan. The project focuses on this group of patients with a less favorable prognosis (with a more aggressive disease). Patients who develop REP within approximately 6 weeks after surgery will have PET/CT (positron emission tomography in combination with computed tomography) examinations using the radiopharmaceutical 11C-methionine in addition to standard practice. PET is one of the most modern methods of molecular imaging, a non-invasive in vivo method that allows physicians to study processes in the human body using radiolabeled radiopharmaceuticals. 11C-methionine is an example of a radiolabeled (carbon 11) amino acid - a source of energy for tumor cells and a building material for new proteins. This radiopharmaceutical is commonly used in the diagnosis of brain tumors and in the evaluation of response to treatment. For patients who undergo this examination, the radiotherapy planning will be adjusted based on it. The purpose of clinical trial is to improve the prospects of patients with REP.

DETAILED DESCRIPTION:
Glioblastoma (GB) is the most aggressive diffuse glioma that corresponds to grade 4 based on the 2016 WHO Classification of Tumors of the Central Nervous System. GB is the most common primary brain malignancy with the incidence of 3 per 100,000 persons per year, accounting for 45 % of malignant primary brain tumors and 54 % of all gliomas. Despite the considerable improvements in surgical techniques, which enable more extensive degree of resection, wide application of more precise radiotherapy (RT) and novel chemotherapeutic agents, GB remains an incurable disease with a median survival of 15 months and 3-year overall survival (OS) of less than 10 % in real clinical practice. Clinical trials evaluating the role of modern targeted therapy did not prove superiority of this treatment strategy and results of GB treatment remains poor.

Current standard of care is based on multimodality treatment combining surgery, RT and chemotherapy with alkylating agent temozolomide (TMZ). Standard post-surgery treatment of newly diagnosed GB patients has remained unchanged since implementation of the recommendations of the EORTC 26981-22981/NCIC CE3 trial (Stupp regimen) that finished enrolling patients in 2002 and was published in 2005. Co-administration of TMZ improved survival from 12,1 months (with RT alone) to 14,6 months (with addition of TMZ). Continuing effort how to improve treatment outcomes is urgent clinical as well as research need.

The phenomenon of postoperative REP has only recently been explored with increasingly available MRI for both postsurgery and preRT indication and is currently of high interest. REP diagnosis is based on a comparison of early postoperative MRI findings (up to 72 hours postoperatively) and planning preRT MRI. Our retrospective analysis of 95 patients with GB treated during 2014-2017 revealed that 52% patients developed suspected progression at MRI performed for RT planning purposes. These patients may represent a subset of patients with a particularly aggressive phenotype of GB. It was consistently confirmed that the presence of early recurrence on planning MRI examination was associated with a more aggressive form of glioblastoma and worse overall survival. Higher risk can be expected in patients after fewer radical resections.

Currently, it is not clear what is the optimal approach in patients with REP. Whether to indicate reoperation of recurrence, to choose accelerated RT regimes with or without concurrent chemotherapy or administration of more aggressive and intensive chemotherapy with combined alkylating cytostatics. Treatment of these patients today is not different from patients without REP, and if so, it is purely an individual approach. Clearly, these patients biased previous clinical trials where no routine preRT MRI examination was performed. Currently, these patients are usually excluded from clinical trials, moreover, recent studies often randomize patients after the competition of standard adjuvant chemoRT without any clear progression on the first post chemoRT MRI. REP in MRI planning is a significant negative prognostic factor that should be a stratification factor in future clinical trials. The basic problem is the postoperative prediction of early recurrence.

Amino acid Carbon-11-labeled methionine PET (MET PET) is the most widely studied tracer for molecular imaging in glioma. PET is currently becoming progressively more established part of brain imaging in both pretreatment as well as follow up examination. There is increasing evidence supporting implementation of PET imaging into brain cancer management. Amino acid tracers´ uptake reflects amino acid transport and proteosynthesis which are increased in most types of tumors including gliomas when compared to normal surrounding tissues. Resulted higher tumor-to-normal brain ratio (T/N ratio) provides higher contrast and tumor discrimination comparing to FDG even through lower absolute standard uptake values (SUV). However, because amino acid tracer transport is independent of blood brain barrier breakdown, there is visible PET uptake for tumors that do not enhance on MRI or for aggressive parts of tumor with no MRI contrast uptake yet.

MET PET plays an especially important role in improving diagnostic procedures for treating brain tumors. [11C] Methionine is not taken up by normal brain tissue to a marked degree, and the sensitivity of MET PET for detecting glioma tumors appears to be high. It has been suggested that MET PET may more precisely outline the true extent of viable tumor tissue than MRI, whereas MRI has the capability to better delineate the total extent of associated pathologic changes, such as edema, in adjacent brain areas. MET PET tumor/normal tissue index of 1,3 was considered the threshold for malignant activity based on correlation to stereotactic histopathology examination. Usage of MET PET is limited by its short half-life to centers with its own cyclotron enabling the manufacture of radiopharmaceuticals. Patients with REP of GB need to start oncological treatment as soon as possible and it is not ethical to wait for other commercially available radiopharmaceuticals (FET, FLT and others) that have a longer half-life but are only available in limited ordering schedule. In the comprehensive neurooncological centers, however, the individual rapid preparation of methionine tracer, the most studied substance in brain tumors, is the unique option how to improve outcomes of patients with REP, particularly aggressive GB.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a person with a histologically proven diagnosis of glioblastoma (GB) according to WHO 2016.
2. The subject is male or female, aged 18 years or older.
3. Performance status (PS) according to ECOG (Eastern Cooperative Oncology Group) 0-2.
4. Healed operation wound.
5. Post-operative MR up to 72 hours.
6. Indication to adjuvant chemoradiotherapy.
7. Patient has to express his/her informed consent and sign the form before the screening period.
8. Detected rapid early progression.
9. Patient must achieve following values of laboratory parameters in the peripheral blood during the screening period:

   1. neutrophiles (total count) ≥1500/mm3
   2. platelets (total count) ≥100 000/mm3
   3. hemoglobin ≥ 9,0 g/dL
   4. serum creatinin ≤1,5x of upper limit of normal, ULN
   5. total bilirubin 1,5x ULN, unless documented Gilbert's syndrome, for which bilirubin ≤ 3x ULN is permitted
   6. AST/ALT ≤3x ULN

Exclusion Criteria:

1. Prior brain surgery.
2. Prior radiotherapy targeting brain.
3. The history of active/currently treated cancer (solid tumor); the exceptions are: non-melanoma skin cancer, in situ bladder carcinoma, in situ gastric cancer, in situ colorectal carcinoma, in situ cervical carcinoma, in situ breast cancer.
4. Any systemic disease or health condition that might posses a risk at anticancer therapy and imaging techniques (MRI, MET PET).
5. Patients must not have substance abuse disorders that would interfere with cooperation with the requirements of the trial.
6. Patients must not have any evidence of ongoing (active) infection (HIV, hepatitis A, B, C).
7. Pregnant and/or breastfeeding women.
8. Patient who disagree and refuses to sign an Informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) in 11C-Methionine PET/CT Arm vs. PFS in Arm Ahist | 44 months
  PFS in 11C-Methionine PET/CT Arm vs. PFS in historical cohort (Arm A/hist./). PFS timeframe = start of radiotherapy / progression of disease or death.

SECONDARY OUTCOMES:
Rapid-Early-Progression incidence | 38 months
  Prospective evaluation of the incidence of Rapid-Early-Progression (REP) on planning MR in patients with GB indicated for adjuvant chemoradiotherapy.
Overall survival in 11C-Methionine PET/CT Arm vs. overall survival in Arm Ahist | 44 months
  OS in 11C-Methionine PET/CT Arm compared to the historical retrospective group (arm Ahist). OS timeframe = surgery / death related to glioblastoma multiforme
Progression free survival in 11C-Methionine PET/CT Arm vs. progression free survival in Arm Ahist. | 44 months
  Median PFS in arm A > median PFS in arm Ahist by ≥3.1 months. Progression free survival (PFS) is defined as the time from initiation of radiotherapy to the occurrence of progression or death.
Biomarkers I | 38 months
  Immunohistochemical analysis of GFAP, Ki-67, IDH1, ATRX, and PDL1. GFAP: positive/negative/focal positive Ki-67, IDH1: positive/negative ATRX loss of expression: positive/negative PDL1 protein expression: positive/negative
Biomarkers II | 38 months
  Mutational status of TERT and IDH2: mutated/wild-type
Biomarkers III | 38 months
  Sanger sequencing of IDH1 in IDH1 IHC positive patients: mutated/wild-type
Biomarkers IV | 38 months
  MGMT promotor methylation status: ≥25% = methylated/<25% = unmethylated
Biomarkers V | 38 months
  1p/19q co-deletion: positive/negative
Patterns-of-failure analysis | 44 months
  Evaluation of spatial patterns of failure (PoF; central (V95% ≥ 95%)/in-field (80% ≤ V95%)/marginal (20% ≤V95% < 80%)/distant (V95% < 20%)) in patients with REP (arm A) compared to the historical retrospective group (arm Ahist). In the case of MULTIFOCAL progression, each PD is evaluated independently, i.e. patient could have one central and one distal PD. In subsequent statistical analysis, each PD is evaluated independently. PoF could be performed even in death subjects, if MR describing the progression is available.
Quality of Life assessment using the standardized European Organisation for Research and Treatment of Cancer (EORTC) questionnaire QLQ-C30 | 44 months
  Quality of life will be assessed using standardized questionnaire: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 v.3.0 during screening period, visits 2, 4, 6, 8, 10, 12 (End-Of-Treatment) and during follow-up period every 3 months (+/- 1 week) up to progression of the disease.
Quality of Life assessment using the standardized European Organisation for Research and Treatment of Cancer (EORTC) Quality of life questionnaire-BN20 | 44 months
  Quality of life will be assessed using standardized questionnaire: additional module Brain cancer European Organisation for Research and Treatment of Cancer Quality of life questionnaire BN20 during screening period, visits 2, 4, 6, 8, 10, 12 (End-Of-Treatment) and during follow-up period every 3 months (+/- 1 week) up to the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Radek Lakomy, MD, Ph.D., Principal Investigator — Masaryk Memorial Cancer Institute, Dept. of Comprehensive Cancer Care
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakomy R, Fadrus P, Slampa P, Svoboda T, Kren L, Lzicarova E, Belanova R, Sikova I, Poprach A, Schneiderova M, Prochazkova M, Sana J, Slaby O, Smrcka M, Vyzula R, Svoboda M. [Multimodal treatment of glioblastoma multiforme: results of 86 consecutive patients diagnosed in period 2003-2009]. Klin Onkol. 2011;24(2):112-20. Czech. PMID 21644366
- [Background] Weller M, van den Bent M, Tonn JC, Stupp R, Preusser M, Cohen-Jonathan-Moyal E, Henriksson R, Le Rhun E, Balana C, Chinot O, Bendszus M, Reijneveld JC, Dhermain F, French P, Marosi C, Watts C, Oberg I, Pilkington G, Baumert BG, Taphoorn MJB, Hegi M, Westphal M, Reifenberger G, Soffietti R, Wick W; European Association for Neuro-Oncology (EANO) Task Force on Gliomas. European Association for Neuro-Oncology (EANO) guideline on the diagnosis and treatment of adult astrocytic and oligodendroglial gliomas. Lancet Oncol. 2017 Jun;18(6):e315-e329. doi: 10.1016/S1470-2045(17)30194-8. Epub 2017 May 5. PMID 28483413
- [Background] Kazda T, Dziacky A, Burkon P, Pospisil P, Slavik M, Rehak Z, Jancalek R, Slampa P, Slaby O, Lakomy R. Radiotherapy of Glioblastoma 15 Years after the Landmark Stupp's Trial: More Controversies than Standards? Radiol Oncol. 2018 Jun 6;52(2):121-128. doi: 10.2478/raon-2018-0023. eCollection 2018 Jun. PMID 30018514
- [Background] Blumenthal DT, Gorlia T, Gilbert MR, Kim MM, Burt Nabors L, Mason WP, Hegi ME, Zhang P, Golfinopoulos V, Perry JR, Hyun Nam D, Erridge SC, Corn BW, Mirimanoff RO, Brown PD, Baumert BG, Mehta MP, van den Bent MJ, Reardon DA, Weller M, Stupp R. Is more better? The impact of extended adjuvant temozolomide in newly diagnosed glioblastoma: a secondary analysis of EORTC and NRG Oncology/RTOG. Neuro Oncol. 2017 Aug 1;19(8):1119-1126. doi: 10.1093/neuonc/nox025. PMID 28371907
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Pirzkall A, McGue C, Saraswathy S, Cha S, Liu R, Vandenberg S, Lamborn KR, Berger MS, Chang SM, Nelson SJ. Tumor regrowth between surgery and initiation of adjuvant therapy in patients with newly diagnosed glioblastoma. Neuro Oncol. 2009 Dec;11(6):842-52. doi: 10.1215/15228517-2009-005. PMID 19229057
- [Background] Wee CW, Kim E, Kim TM, Park CK, Kim JW, Choi SH, Yoo RE, Lee ST, Kim IH. Impact of interim progression during the surgery-to-radiotherapy interval and its predictors in glioblastoma treated with temozolomide-based radiochemotherapy. J Neurooncol. 2017 Aug;134(1):169-175. doi: 10.1007/s11060-017-2505-x. Epub 2017 May 25. PMID 28547592
- [Background] Merkel A, Soeldner D, Wendl C, Urkan D, Kuramatsu JB, Seliger C, Proescholdt M, Eyupoglu IY, Hau P, Uhl M. Early postoperative tumor progression predicts clinical outcome in glioblastoma-implication for clinical trials. J Neurooncol. 2017 Apr;132(2):249-254. doi: 10.1007/s11060-016-2362-z. Epub 2017 Jan 18. PMID 28101701
- [Background] Katsanos AH, Alexiou GA, Fotopoulos AD, Jabbour P, Kyritsis AP, Sioka C. Performance of 18F-FDG, 11C-Methionine, and 18F-FET PET for Glioma Grading: A Meta-analysis. Clin Nucl Med. 2019 Nov;44(11):864-869. doi: 10.1097/RLU.0000000000002654. PMID 31205150
- [Background] Grosu AL, Weber WA, Riedel E, Jeremic B, Nieder C, Franz M, Gumprecht H, Jaeger R, Schwaiger M, Molls M. L-(methyl-11C) methionine positron emission tomography for target delineation in resected high-grade gliomas before radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):64-74. doi: 10.1016/j.ijrobp.2005.01.045. PMID 16111573
- [Background] Matsuo M, Miwa K, Tanaka O, Shinoda J, Nishibori H, Tsuge Y, Yano H, Iwama T, Hayashi S, Hoshi H, Yamada J, Kanematsu M, Aoyama H. Impact of [11C]methionine positron emission tomography for target definition of glioblastoma multiforme in radiation therapy planning. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):83-9. doi: 10.1016/j.ijrobp.2010.09.020. Epub 2010 Nov 20. PMID 21095072
- [Derived] Lakomy R, Lojova M, Souckova L, Hynkova L, Polachova K, Vasina J, Demlova R, Poprach A, Sana J, Prochazka T, Smrcka M, Fadrus P, Jancalek R, Selingerova I, Belanova R, Slampa P, Pospisil P, Kazda T. 11C-methionine in the diagnostics and management of glioblastoma patients with rapid early progression: nonrandomized, open label, prospective clinical trial (GlioMET). BMC Cancer. 2024 Jun 15;24(1):736. doi: 10.1186/s12885-024-12469-2. PMID 38879476